CLINICAL TRIAL: NCT01963065
Title: Chemical Exposures and Infant Outcomes in the Neonatal Intensive Care Unit
Brief Title: NICU-HEALTH (Hospital Exposures and Long-Term Health)
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Annemarie Stroustrup, Principal Investigator, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 12-0332; 1K23ES022268-01 (NIH)
Record Dates: First submitted 2013-09-24; First posted 2013-10-16 (Estimated); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Preterm Birth
Keywords: Children's environmental health; Preterm birth; Newborns; Bisphenol A; BPA; Phthalates; Metals exposure; Very low birth weight; NICU; Stress
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with DNA - samples retained, with potential for extraction of DNA from at least one fo the types of samples retained (e.g., frozen tissue, whole blood)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Moderately pre-term infants and their mothers: cohort of moderately pre-term infants and their mothers

SUMMARY:
The purpose of this study is to evaluate the impact of environmental exposures during the NICU hospitalization on preterm infant development. The research team is interested in both chemical and non-chemical exposures. Research studies have shown that babies are exposed to plasticizers (bisphenol A, phthalates) in the NICU. Plasticizers are chemicals that are used to make plastic medical equipment soft and flexible. The research team wants to find out whether NICU-based exposure to chemicals (including common plasticizers) and other non-chemical exposures like stress makes a difference to how they grow and develop.

DETAILED DESCRIPTION:
1. Significance Premature newborns may be particularly vulnerable to the effects of toxic chemicals in the environment because of their small body size, immature hepatic and renal clearance mechanisms, and rapid rate of development. Approximately 8% of neonates in the United States require admission to a NICU following birth; thus over 300,000 infants annually are exposed to the chemical-intensive hospital environment during a developmentally vulnerable period. Infants cared for in the NICU have increased risk of developmental delay, cognitive dysfunction, attention deficit hyperactivity disorder, and autism that is only partially explained by degree of prematurity or severity of clinical disease. Abnormalities found on neuroimaging are relatively insensitive predictors of long-term cognitive and behavioral outcome. Moreover, many medical conditions associated with prematurity, such as chronic lung disease and retinopathy of prematurity, are incompletely predicted by gestational age at birth or severity of newborn illness. The study team hypothesizes that a portion of the neurocognitive, social, and somatic impairments seen in NICU graduates are attributable to potentially preventable NICU-based exposures.

   As NICU care has matured, survival is likely for all but the most premature infants. The research emphasis is therefore shifting from survival to developing methods for improving the long term growth and development of the patients. The study team believes this research strategy must examine the potential contribution of environmental exposures that occur during the NICU stay as predictors of outcome. All subjects in the proposed study are cared for in the NICU - therefore comparisons are internally valid. While findings may not be generalizable to non-NICU populations, the potential positive impact of this work on thousands of NICU graduates makes this work a high impact public health priority. The study team's focus moderately premature infants as these infants generally experience much of the third trimester developmental window ex utero in the NICU, but generally have low rates of significant disease related to prematurity (such as intraventricular hemorrhage, bronchopulmonary dysplasia, etc). Studies of in utero exposure to common environmental chemicals and stress indicate the vulnerability of developmentally immature individuals during this same developmental window. It is therefore logical to assess whether ex utero exposures occurring in the NICU act similarly. Additionally, small cross-sectional studies indicate the high exposure levels faced by NICU inpatients. Through this study, the study team's plan to characterize the role of hospital-based exposures on preterm infant development.
2. Preliminary Studies and Innovation: Substantial information on the health effects of community-based early life exposure, as well as the presence in the NICU environment, exist for both stress and the chemicals of interest in this study. Numerous materials used in NICU care, such as incubators, respiratory support devices, and intravenous (IV) and enteral feeding supplies, are made from plastics that act as vehicles of chemical exposure. Phthalates - chemicals used to make plastic flexible and resilient - are common in medical materials. Bisphenol A (BPA) and other organic phenols, as well as contaminating metals are also present in plastic materials. Silver is added to plastic IV catheter components as an antimicrobial. Parenteral nutrition (PN), frequently administered for long duration in the NICU, contains Mn. Surprisingly, there is little evidence to support the safety of the total dose of Mn added to PN, and a growing body of literature suggests that Mn toxicity may be occurring among NICU patients. Exposure to these chemicals may be associated with significant developmental impairment, however, the impact of early-life chemical exposure on neurodevelopment in NICU graduates is largely unstudied.
3. Evolving evidence suggests that chemical and non-chemical stressors in the NICU may impact infant neurodevelopment. The built environment, ambient noise, in-hospital parent-child interactions, and parental stress during the NICU stay have been associated with altered neurodevelopment among NICU graduates. Socioeconomic factors and psychological functioning of the primary caregiver are also linked to childhood neurodevelopmental outcomes generally. These factors must therefore be considered as confounders and/or modifiers in any comprehensive NICU neurodevelopmental outcome association study.
4. Study Goals and Plan: This study will identify specific sources of chemical exposure among NICU inpatients and explore the association between exposure and outcomes. It will also measure biomarkers of stress response and evaluate the relationship between stress and outcome. The proposed study will identify the prevalence and dose of chemicals to which NICU inpatients are exposed and provide data on associations with neurodevelopmental outcomes. The study team has picked a small number of candidate chemicals for which exposure is known or likely, the negative neurodevelopmental impact of community exposure is documented, and the health implications for NICU-based exposure are unknown. Prior studies have documented numerous phthalate-containing materials in the NICU and elevated biomarkers of phthalates and BPA in NICU inpatients. These studies were limited by cross-sectional specimen sampling, patient enrollment without attention to factors likely to affect chemical metabolism including gestational or chronologic age and severity of illness, and small sample size. To the study team's knowledge, biomarkers of NICU-exposure to Ag, Cd, and Mn have not been assessed, despite the documented presence of these metals in the NICU and known adverse health outcomes related to early life exposure. No previous study of NICU chemical exposure has considered the important potential confounders/modifiers of chemical toxicant impact to be considered in the proposed study. No rigorous study has evaluated biomarkers of stress and association with outcomes in the NICU hospitalization.

The relationship between biomarkers of exposure to chemicals in the NICU and specific care practices has not been explored previously. Additionally, the potential association between NICU-based chemical or stress exposures and neurodevelopmental deficits has not been evaluated. Two previous studies assessed outcomes related to NICU phthalate exposure, but neither used exposure biomarkers or other validated exposure assessment methods to characterize initial exposure nor considered important non-chemical confounders.

The NICU-HEALTH cohort addresses these limitations and is a comprehensive, longitudinal evaluation of chemical exposure in the NICU designed to evaluate environmental chemical exposure and clinical outcomes in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Birth at Mount Sinai Hospital
* Gestational age at birth 28-0/7 through 32-6/7 weeks

Exclusion Criteria:

* Birth at an outside hospital
* Chromosomal abnormality or other genetic disorder
* Concern for hypoxic-ischemic encephalopathy
* Inborn error of metabolism
* Congenital renal disease
* Intestinal obstruction
* Major congenital anomaly

Max Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Neonates born 28-0/7 through 32-6/7 weeks gestation admitted to the Mount Sinai NICU are be eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-04-28 (Actual)

PRIMARY OUTCOMES:
NICU Network Neurobehavioral Scale | at 34-42 weeks postmenstrual age
  Performance on a scale of newborn neurodevelopment designed both for use in newborns exposed to toxins in utero and for evaluation of infants born preterm

SECONDARY OUTCOMES:
Dense-array electroencephalogram | at 34-42 weeks postmenstrual age
  Dense-array EEG is a measure of infant neurologic function. The use of commercially-available high-density array mesh caps (Electrical Geodesics, Inc., Eugene, OR) allows the EEG to be placed on a study subject in under five minutes, and is comfortable enough to remain in place through multiple care activities and during sleep. Dense-array EEG has been used successfully used to demonstrate varying electrocortical functional connectivity between babies born at term or preterm, and has been correlated to performance on neurocognitive tests later in life.

CONTACTS AND LOCATIONS:
Overall Officials: Annemarie Stroustrup, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Stroustrup A, Bragg JB, Busgang SA, Andra SS, Curtin P, Spear EA, Just AC, Arora M, Gennings C. Sources of clinically significant neonatal intensive care unit phthalate exposure. J Expo Sci Environ Epidemiol. 2020 Jan;30(1):137-148. doi: 10.1038/s41370-018-0069-2. Epub 2018 Sep 21. PMID 30242269
- [Background] Stroustrup A, Bragg JB, Andra SS, Curtin PC, Spear EA, Sison DB, Just AC, Arora M, Gennings C. Neonatal intensive care unit phthalate exposure and preterm infant neurobehavioral performance. PLoS One. 2018 Mar 5;13(3):e0193835. doi: 10.1371/journal.pone.0193835. eCollection 2018. PMID 29505594
- [Background] Stroustrup A, Teitelbaum SL, Aschner JL. The Value of Preterm Infant Environmental Health Cohorts: The Canary in the Coal Mine. JAMA Pediatr. 2017 Dec 1;171(12):1139-1140. doi: 10.1001/jamapediatrics.2017.3230. No abstract available. PMID 29059271
- [Background] Stroustrup A, Bragg JB, Spear EA, Aguiar A, Zimmerman E, Isler JR, Busgang SA, Curtin PC, Gennings C, Andra SS, Arora M. Cohort profile: the Neonatal Intensive Care Unit Hospital Exposures and Long-Term Health (NICU-HEALTH) cohort, a prospective preterm birth cohort in New York City. BMJ Open. 2019 Nov 25;9(11):e032758. doi: 10.1136/bmjopen-2019-032758. PMID 31772104